CLINICAL TRIAL: NCT03893435
Title: The Role of Sacubitril/Valsartan in Post-acute Myocardial Infarction: The RSVP-AMI Trial
Brief Title: The Role of Sacubitril/Valsartan in Post-acute Myocardial Infarction
Acronym: RSVP-AMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Young Investigator Group of Cardiovascular Research (Network)
Responsible Party: Principal Investigator, Abdallah Almaghraby, Senior Registrar of Cardiology and Angiology, The Young Investigator Group of Cardiovascular Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YIG01201902
Record Dates: First submitted 2019-03-10; First posted 2019-03-28 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — sacubitril; Valsartan; sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacubitril/Valsartan (Experimental): In successfully revascularized post-AMI patients with LVEF ≤40% Sacubitril/Valsartan with the recommended starting dose: 24 mg/26 mg PO BID. After 2-4 weeks, the dose will be doubled to the target maintenance dose of 97 mg/103 mg PO BID (if tolerated) for 6 months.
  Interventions: Drug: Sacubitril / Valsartan Oral Tablet [Entresto]
- Valsartan (Active Comparator): In successfully revascularized post-AMI patients with LVEF ≤40% Valsartan with an initial dose of 40 mg PO BID, with subsequent titrations to target maintenance dose of 160 mg BID as tolerated.
  Interventions: Drug: Sacubitril / Valsartan Oral Tablet [Entresto]

INTERVENTIONS:
Drug: Sacubitril / Valsartan Oral Tablet [Entresto] — Sacubitril/Valsartan with the recommended starting dose: 24 mg/26 mg PO BID. After 2-4 weeks, the dose will be doubled to the target maintenance dose of 97 mg/103 mg PO BID (if tolerated) for 6 months.
  Other Names: ARNI

SUMMARY:
Sacubitril/Valsartan (SAC/VAL) is a new treatment of congestive heart failure (CHF) recently indicated as class I, level of evidence B in the recent European Society of Cardiology (ESC) guidelines 2016 of CHF. PARADIGM-HF trial demonstrated a significant improvement of morbidity and mortality with SAC/VAL in comparison to enalapril. So far, no data available about the effect of usage of SAC/VAL post-acute myocardial infarction (AMI) except in animal experimental models.

The purpose of the research is evaluation of the effects of SAC/VAL in post-AMI in comparison to the traditional Angiotensin Converting Enzyme inhibitors (ACEs inhibitors) or Angiotensin II Receptor Blockers (ARBs) in a real-life clinical trial in treatment of post-AMI patients with reduced left ventricular (LV) systolic function.

DETAILED DESCRIPTION:
Background and study rationale:

Sacubitril/Valsartan (SAC/VAL) is now approved by the U.S. Food and Drug Administration (FDA) for heart failure with reduced ejection fraction (HFrEF) and also, recently indicated as class I indication, level of evidence B in the European Society of Cardiology (ESC) guidelines 2016 on congestive heart failure (CHF).(1) PARADIGM-HF trial demonstrated that morbidity and mortality can be improved with SAC/VAL In comparison to enalapril, it reduced the occurrence of cardiovascular death or hospitalization for CHF by 20% with a 16% reduction in all-cause mortality.(2) So far, no available data about the effect of usage of SAC/VAL in post-AMI except in animal experimental models that proved efficacy of SAC/VAL in preventing AMI-induced LV dysfunction compared with SAC/VAL, also significantly attenuated LV scar size following AMI compared with placebo .(3)

Aim of the work:

* This study aims to investigate the effects of SAC/VAL in post-AMI through using it instead of conventional Angiotensin Converting enzyme inhibitors (ACEs inhibitors) or Angiotensin II Receptor Blockers (ARBs) in treatment of post-AMI patients with reduced left ventricular (LV) systolic function.
* Design: Randomized open label interventional clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Post-AMI patients who underwent successful PPCI and LVEF ≤40%.

Exclusion Criteria:

* Post-AMI patients who underwent successful PPCI and LVEF >40%.
* History of hypersensitivity or allergy to any of the study drugs, as well as known or suspected contraindications to the study drugs.
* Symptomatic hypotension and/or an SBP < 100 mmHg.
* Estimated GFR < 30 mL/min/1.73m2 as measured by the simplified MDRD formula or serum potassium > 5.2 mmol/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
One week major adverse cerebrovascular and cardiovascular events (MACCE) | 1 week after AMI
  Major adverse cerebrovascular and cardiovascular events (MACCE) will be assessed 1 week after AMI
Twenty four weeks major adverse cerebrovascular and cardiovascular events (MACCE) | 24 weeks after AMI
  Major adverse cerebrovascular and cardiovascular events (MACCE) will be assessed 24 weeks after AMI
Change in the ejection fraction during hospital stay, 3 months and 6 months after AMI. | In hospital, 3 months and 6 months after AMI
  Change in the ejection fraction assessed by transthoracic echocardiography assessment (TTE) during hospital stay, 3 months and 6 months after AMI.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif S Elbeltagui, MD, Study Director — Assisstant Professor of Cardiology, University of Alexandria, Egypt
Locations (1):
- Andalusia Hospitals, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No